CLINICAL TRIAL: NCT00091195
Title: A Phase II Study Of Single Agent Depsipeptide (FK228) In Recurrent, Platinum Sensitive Adeno-Carcinoma Of The Ovary Or Peritoneum
Brief Title: Depsipeptide (Romidepsin) in Treating Patients With Recurrent Ovarian Epithelial or Peritoneal Cavity Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01036; CCCWFU 83403; U10CA081851 (NIH); NCT01645670 (obsolete NCT alias); NCT01660282 (obsolete NCT alias)
Record Dates: First submitted 2004-09-07; First posted 2004-09-09 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — romidepsin

ARMS (1):
- Treatment (single-agent depsipeptide) (Experimental): Patients receive depsipeptide (romidepsin) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: romidepsin

INTERVENTIONS:
Drug: romidepsin
  Other Names: FK228; FR901228; Istodax

SUMMARY:
This phase II trial is studying how well depsipeptide (romidepsin) works in treating patients with recurrent ovarian epithelial or peritoneal cavity cancer. Drugs used in chemotherapy, such as depsipeptide (romidepsin), work in different ways to stop tumor cells from dividing so they stop growing or die. Depsipeptide (romidepsin) may also stop the growth of ovarian epithelial or peritoneal cavity cancer by stopping blood flow to the tumor and by blocking the enzymes necessary for their growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the response rate of recurrent, platinum-sensitive adenocarcinoma of the ovarian or peritoneal to depsipeptide (romidepsin).

II. To determine the toxicity of depsipeptide in this patient population.

OUTLINE: This is a multicenter study.

Patients receive depsipeptide (romidepsin) intravenously (IV) over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed primary ovarian epithelial or peritoneal cavity cancer

  * Histologic confirmation of recurrent disease not required
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques (including palpation, plain x-ray, computed tomography [CT] scan, or magnetic resonance imaging [MRI]) OR ≥ 10 mm by spiral CT scan
* Achieved a complete response after initial prior platinum-containing (cisplatin or carboplatin) chemotherapy regimen (e.g., conventional-dose therapy, high-dose therapy, consolidation therapy, or extended therapy after surgical or nonsurgical assessment)

  * Patients who have not received paclitaxel or docetaxel as initial therapy may receive a second regimen containing these drugs
  * No prior chemotherapy for persistent or recurrent disease, including re-treatment with the original regimen
* Platinum-sensitive disease, defined as having a treatment-free interval with no evidence of progressive disease for > 6 but < 12 months after completion of a platinum-based regimen
* No known brain metastases
* Performance status - Eastern Cooperative Oncology Group (ECOG) 0-2
* Performance status - Karnofsky 60-100%
* More than 6 months
* White blood cells (WBC) ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* Creatinine clearance ≥ 60 mL/min
* No New York Heart Association class III or IV congestive heart failure
* No myocardial infarction within the past year
* No uncontrolled dysrhythmias
* No poorly controlled angina
* No history of serious ventricular arrhythmia (e.g., ventricular tachycardia or ventricular fibrillation, ≥ 3 beats in a row)
* QTc interval < 500 msec
* No other significant cardiac disease
* Potassium normal
* Magnesium normal
* No uncontrolled electrolyte abnormality (hypokalemia and hypomagnesemia)
* No ongoing or active infection requiring antibiotics
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to study drug
* No neuropathy ≥ grade 2
* No other uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior monoclonal antibodies, cytokines, or signal transduction inhibitors for recurrent disease
* No concurrent biologic therapy
* See Disease Characteristics
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) for the primary malignancy
* No prior FR901228 (depsipeptide)
* No other concurrent chemotherapy
* More than 4 weeks since prior hormonal therapy for the primary malignancy
* Concurrent estrogen replacement therapy allowed
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to > 25% of bone marrow
* No concurrent radiotherapy
* Recovered from all prior therapy
* More than 4 weeks since prior noncytotoxic therapy for the primary malignancy
* No other prior noncytotoxic therapy for recurrent disease
* No concurrent combination anti-retroviral therapy for HIV-positive patients
* No other concurrent drugs known to have histone deacetylase inhibitor activity (e.g., valproic acid)
* No concurrent agents that cause QTc prolongation
* No other concurrent investigational agents
* No other concurrent anticancer agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2004-09; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 5 years
  Estimated as proportion of patients with complete or partial reduction in tumor burden.
Toxicity as assessed by CTCAE version 3.0 | Up to 5 years
Time to progression | From first treatment until the date of progression, assessed up to 5 years
Survival | From first treatment until death or the last date of contact, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Miller, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - High Point Regional Hospital, High Point, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina